CLINICAL TRIAL: NCT05225207
Title: A Study of Lenvatinib in Korean Unresectable Hepatocellular Carcinoma (uHCC) Patients as a Post-marketing Surveillance
Brief Title: A Study of Lenvima (Lenvatinib) in Korean Unresectable Hepatocellular Carcinoma (uHCC) Participants
Status: Completed | Type: Observational
Sponsor: Eisai Korea Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: E7080-M082-509
Record Dates: First submitted 2022-01-26; First posted 2022-02-04 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-01

CONDITIONS: Liver Neoplasms; Carcinoma, Hepatocellular
Keywords: Lenvatinib; Lenvima
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All Participants: Participants with uHCC who are prescribed with Lenvima within the scope of the approved label for Korea under the medical judgment of the investigator will be enrolled and observed for up to 12 months.
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — No intervention will be administered.

SUMMARY:
The purpose of this study is to describe the following safety and the efficacy of Lenvima for the first-line treatment indication of participants with uHHC in the post marketing setting: (1) Serious adverse events and serious adverse drug reactions (2) Unexpected adverse events and adverse drug reactions not reflected in the precautions for use (3) Known adverse drug reactions (4) Non-serious adverse drug reactions (5) Other safety and efficacy related information.

ELIGIBILITY:
Inclusion Criteria:

1. Participants over 18 years
2. Participants who are treated with lenvatinib according to the approved indication of uHCC as first-line therapy in Korea
3. Participants who have given their consent to study participation about the use of the personal data and medical data

Exclusion Criteria:

1. Participants who have hypersensitivity to active pharmaceutical ingredients or excipient of the study drug (lenvatinib)
2. Participants who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with uHHC administered with Lenvima within the scope of the approved label for Korea under the medical judgment of the investigator.
Sampling Method: Non-Probability Sample
Enrollment: 658 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Serious Adverse Events (SAEs) | From first dose of study drug up to 12 months
  A SAE is defined as any untoward medical occurrence: resulting in death; life threatening requiring hospitalization or prolongation of hospitalization; resulting in persistent or significant disability or incapacity; resulting in birth defect or congenital anomaly or medically important due to other reasons than above mentioned criteria.
Number of Participants With Serious Adverse Drug Reactions (ADRs) | From first dose of study drug up to 12 months
  Serious ADR is defined as any untoward medical occurrence or effect that at any dose resulted in death or life-threatening conditions or required hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, congenital anomaly or birth defect or medically important condition.
Number of Participants With Unexpected AEs | From first dose of study drug up to 12 months
  AE is defined as any untoward and unintended signs (example, anomalies in laboratory test results) or symptoms/diseases occurring during administration/use of drugs, etc., which do not necessarily have a causal relationship with the drug in question.
Number of Participants With Unexpected ADRs | From first dose of study drug up to 12 months
  An ADR is defined as harmful and unintended responses to the normal administration/use of drugs, in which a causal relationship with the drug in question cannot be ruled out. AEs with unknown causality to the drug among those voluntarily reported will be also considered ADRs.
Number of Participants With Known ADRs | From first dose of study drug up to 12 months
  An ADR is defined as harmful and unintended responses to the normal administration/use of drugs, in which a causal relationship with the drug in question cannot be ruled out. AEs with unknown causality to the drug among those voluntarily reported will be also considered ADRs.
Number of Participants With Non-serious ADRs | From first dose of study drug up to 12 months
  An ADR is defined as harmful and unintended responses to the normal administration/use of drugs, in which a causal relationship with the drug in question cannot be ruled out. AEs with unknown causality to the drug among those voluntarily reported will be also considered ADRs.

SECONDARY OUTCOMES:
Percentage of Participants With Overall Response | From first dose of study drug up to 12 months
  Overall response will include complete response (CR), and partial response (PR). The confirmation of overall response will be based on investigator's judgement.

CONTACTS AND LOCATIONS:
Locations (42):
- South Korea (42):
  - Site #32, Cheonan, Chungcheongnam-do
  - Site #35, Bucheon-si, Gyeonggi-do
  - Site #38, Bucheon-si, Gyeonggi-do
  - Site #06, Goyang-si, Gyeonggi-do
  - Site #03, Seongnam-si, Gyeonggi-do
  - Site #13, Suwon, Gyeonggi-do
  - Site #27, Suwon, Gyeonggi-do
  - Site #15, Uijeongbu-si, Gyeonggi-do
  - Site #37, Changwon, Gyeongsangnam-do
  - Site #28, Yangsan, Gyeongsangnam-do
  - Site #29, Yangsan, Gyeongsangnam-do
  - Site #31, Busan
  - Site #39, Busan
  - Site #40, Busan
  - Site #17, Daegu
  - Site #18, Daegu
  - Site #26, Daegu
  - Site #30, Daegu
  - Site #41, Daegu
  - Site #19, Daejeon
  - Site #20, Daejeon
  - Site #24, Daejeon
  - Site #34, Daejeon
  - Site #21, Incheon
  - Site #33, Incheon
  - Site #36, Incheon
  - Site #01, Seoul
  - Site #02, Seoul
  - Site #04, Seoul
  - Site #07, Seoul
  - Site #08, Seoul
  - Site #09, Seoul
  - Site #10, Seoul
  - Site #12, Seoul
  - Site #16, Seoul
  - Site #22, Seoul
  - Site #23, Seoul
  - Site #25, Seoul
  - Site #42, Seoul
  - Site #43, Seoul
  - Site #44, Seoul
  - Site #11, Ulsan

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.

REFERENCES:
- [Derived] Kang W, Kim YJ, Kim SU, Seo YS, Kim JW, Kim JH, Park SY, Baek YH, Kim KM, Lee HL, Yoon KT, Kim H, Cheong JY, Hwang JS, Kim JH, Kim KM, Sung PS, Kim J, Kim DY. Real-world safety and effectiveness of lenvatinib in unresectable hepatocellular carcinoma in Korea: post-marketing study. Future Oncol. 2024;20(37):2949-2959. doi: 10.1080/14796694.2024.2397328. Epub 2024 Sep 25. PMID 39320906